CLINICAL TRIAL: NCT00002552
Title: AUTOLOGOUS, ALLOGENEIC, OR SYNGENEIC BONE MARROW TRANSPLANTATION IN HODGKIN'S DISEASE, NON-HODGKIN'S LYMPHOMA, AND MULTIPLE MYELOMA
Brief Title: Chemotherapy Plus Bone Marrow Transplantation in Treating Patients With Refractory Non-Hodgkin's Lymphoma, Hodgkin's Disease, or Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000063370; P30CA022453 (NIH); WSU-D-701-87; NCI-V94-0364
Record Dates: First submitted 1999-11-01; First posted 2004-05-24 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm
Keywords: recurrent adult Hodgkin lymphoma; refractory multiple myeloma; recurrent small lymphocytic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult unfavorable prognosis Hodgkin lymphoma; childhood unfavorable prognosis Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Filgrastim; sargramostim; Carmustine; Cyclophosphamide; Cytarabine; Etoposide; Leucovorin; Methotrexate; perfosfamide; Hydrocortisone; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Biological: sargramostim
Drug: carmustine
Drug: cyclophosphamide
Drug: cytarabine
Drug: etoposide
Drug: leucovorin calcium
Drug: methotrexate
Drug: perfosfamide
Drug: therapeutic hydrocortisone
Procedure: allogeneic bone marrow transplantation
Procedure: autologous bone marrow transplantation
Procedure: in vitro-treated bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Procedure: syngeneic bone marrow transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining bone marrow transplantation with chemotherapy may allow doctors to give higher doses of chemotherapy and kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects of giving a bone marrow transplant together with chemotherapy and to see how well it works in treating patients with refractory non-Hodgkin's lymphoma, Hodgkin's lymphoma, or multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the toxicities, response rate, and duration of response associated with high-dose cyclophosphamide, etoposide, carmustine or high-dose cyclophosphamide and total-body irradiation followed by autologous, allogeneic, or syngeneic bone marrow transplant in patients with refractory or high-risk non-Hodgkin's lymphoma, Hodgkin's disease, or multiple myeloma. II. Evaluate any prognostic factors.

OUTLINE: Patients with prior radiotherapy (greater than 2,000 cGy) receive cyclophosphamide IV over 2 hours and etoposide IV over at least 30 minutes on days -7 through -4 followed by carmustine IV over 2 hours on day -3. Patients receive allogeneic or autologous bone marrow transplantation on day 0. Patients with or without prior radiotherapy (less than 2,000 cGy) receive cyclophosphamide IV over 2 hours on days -8 through -5 followed by total body irradiation on days -4 through -1. Patients receive allogeneic or autologous bone marrow transplantation on day 0. Prior to autologous bone marrow transplantation and following myeloablative chemotherapy, patients undergo mobilization consisting of cytarabine subcutaneously every 12 hours for 6 doses. Approximately 24 hours later, patients receive sargramostim (GM-CSF) subcutaneously. Peripheral blood stem cells are collected every 1-3 days beginning when blood counts recover and continuing until sufficient number of cells are reached.

PROJECTED ACCRUAL: Approximately 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven Hodgkin's disease (HD), non-Hodgkin's lymphoma (NHL), and multiple myeloma (MM) meeting the following requirements: Refractory to or at high risk following prior therapy Responded with at least a partial response to last cytoreductive regimen No bulky disease (individual tumor diameter larger than 5 cm) Eligible HD: CNS involvement at original presentation and currently in complete response (CR) Relapsed within 1 year following completion of front-line MOPP or ABVD Relapsed at any time following front-line MOPP/ABVD or other hybrid Eligible NHL: Any grade lymphoma with CNS involvement at original presentation and currently in CR High-grade lymphomas (International Working Formulation H-J) with marrow involvement at original presentation and currently in CR, EXCEPT: Immunoblastic lymphoma and large cell (IWF G and H) with bone marrow involvement with small cleaved cell at original presentation High-/intermediate-grade lymphomas (IWF D-J) in relapse after adequate front-line therapy High-/intermediate-grade lymphomas (IWF D-J) that failed to achieve CR with adequate front-line therapy Low-grade lymphomas (IWF A-C) with B symptoms at original presentation and relapse after front-line therapy Low-grade lymphomas (IWF A-C) in relapse within 1 year following last chemotherapy Low-grade lymphomas (IWF A-C) with documented histologic conversion Eligible MM: Diagnosis based on either presence of both Group I diagnostic criteria OR One Group I criterion and all Group II criteria Group I diagnostic criteria: Plasma cells and/or myeloma cells greater than 10% in bone marrow Biopsy-proven plasmacytoma in bone or soft tissue Group II diagnostic criteria: Monoclonal serum protein spike Urinary myeloma protein Osteolytic lesions on radiologic examination Generalized osteoporosis suffices if plasma cells in marrow exceed 30% Myeloma cells in at least 2 peripheral blood smears Stage II/III disease documented sometime during clinical course Stage III defined by presence of at least 1 of the following: Hemoglobin less than 8.5 g/dl Serum calcium greater than 12 mg/dl Advanced lytic bone lesions High M-component production rates: IgG greater than 7 g/dl IgA greater than 5 g/dl Urinary light chain greater than 4 g/24 hours Stage II disease defined by absence of Stage III characteristics but presence of at least 1 of the following: Hb less than 10 g/dl More than 1 osteolytic lesion, none advanced IgG greater than 5 g/dl IgA greater than 3 g/dl Bone marrow donor available for lymphoma patients with marrow involvement Perfosfamide-purged autologous transplant allowed in patients with no matched sibling donor if: Marrow involvement is limited (less than 30% tumor cells on smears and in bilateral iliac crest biopsies) AND Age is under 60 Donor requirements: Excellent physical condition by history, lab studies, PE No physiologic, psychologic, or medical inability to tolerate the procedure No increased anesthetic risk No HIV infection Priority of multiple donors (in order given): ABO compatible Age over 18 Same sex as recipient A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: 70 and under Performance status: 0-2 Life expectancy: No severe limitation due to nonmalignant disease Hematopoietic: Not specified Hepatic: No severe hepatic disease Bilirubin no greater than 2.0 mg/dL Transaminases no greater than 3 times normal Renal: No severe renal disease Creatinine no greater than 1.5 mg/dL Creatinine clearance at least 60 mL/min Cardiovascular: No symptomatic cardiac disease LVEF at least 50% Pulmonary: No severe pulmonary disease FEV1 and FVC at least 75% of normal Other: No history of severe cystitis with cyclophosphamide No HIV infection No severe personality disorder or severe mental illness No other condition that would markedly increase the morbidity and mortality of transplantation (e.g., substance abuse) Patients with borderline parameters of organ function, performance status, or mental status are entered at the discretion of the transplant team

PRIOR CONCURRENT THERAPY: See Disease Characteristics

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1993-10; Primary Completion 2001-09 (Actual); Study Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Dansey, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States